CLINICAL TRIAL: NCT05307289
Title: Study of Alterations in Tumor Metabolism Associated With the Development of Immunotherapy Resistance in Melanoma
Acronym: MEL-META
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-PP-20
Record Dates: First submitted 2022-03-10; First posted 2022-04-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- melanoma inclusion (Other): Biopsy of a metastasis allowing melanoma diagnosis and realization of primary cultures for metabolomics. An additional 20ml blood sample will also be taken to quantify circulating metabolites and to isolate PBMC.
  Interventions: Other: Biposy

INTERVENTIONS:
Other: Biposy — Biopsy at inclusion visit and at disease progression if applicable

SUMMARY:
Among the mechanisms responsible for resistance to immunotherapy, metabolism seems to play a major role. A better understanding of tumor metabolism appears to be absolutely necessary in order to propose efficient therapeutic alternatives to target tumor cells without exerting a deleterious effect on the cells responsible for the anti-tumor immune response. The main objective is to evaluate metabolism modulations in melanoma cells extracted from metastases of patients sensitive and resistant to immunotherapies (anti-PD1 or anti-PD1+anti-CTLA4).

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18 years of age or older
* Stage III unresectable or histologically confirmed stage IV cutaneous melanoma (melanoma of unknown origin is accepted), treatment naïve (metastatic stage) and for which immunotherapy will be started
* Performance Status ≤1
* BRAF status available; BRAF status determination is required but patient will be eligible regardless of BRAF status
* For women of childbearing potential, effective contraception must be initiated during the study.
* Patient affiliated to social security plan
* Patient having signed informed consent

Exclusion Criteria:

* Breastfeeding or pregnant patients: for women of childbearing age, a urine pregnancy test will be performed
* Patients with ocular or mucosal melanoma of metastatic ocular melanoma
* Patients with metastatic melanoma not treated with immunotherapy (i.e. treated with a combination of targeted therapies).
* Contraindication to the initiation of immunotherapy: HIV and/or HCV and/or HBV positive, active autoimmune disease (chronic inflammatory bowel disease such as ulcerative colitis, Crohn's disease, vasculitis, etc.), patients with autoimmune motor neuropathy (such as Guillain Barré syndrome).
* Vulnerable patients: minors, adults under guardianship or curatorship, deprived of liberty
* Vulnerable persons (minors, patients under guardianship or curatorship, deprived of liberty, under court protection, etc.).
* A psychiatric or addiction history that will compromise the patient's ability to consent and follow the proper protocol procedures
* Any other clinical finding that, in the opinion of the principal investigator, could interfere with the results of the study or pose a risk to the patient during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2028-05-25 (Estimated); Study Completion 2028-10-25 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pyrimidine metabolism at 4 years | At inclusion visit and 4 years
  Investigation of modulations of pyrimidine metabolism using isotopically labelled glutamine

SECONDARY OUTCOMES:
Overall Survival | At inclusion visit and 4 years
  Overall survival (OS) will be measured using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Montaudie Henri, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No